CLINICAL TRIAL: NCT00000246
Title: Rapid Benzodiazepine Detoxification Using Flumazenil
Brief Title: Rapid Benzodiazepine Detoxification Using Flumazenil - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-08265-1; R01DA008265 (NIH); R01-08265-1; NCT00000247 (obsolete NCT alias)
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Substance-Related Disorders
Keywords: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Flumazenil

INTERVENTIONS:
Drug: Flumazenil

SUMMARY:
The purpose of this study is to verify the hypothesis that the benzodiazepine antagonist, flumazenil, will reduce acute benzodiazepine withdrawal.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1993-01; Primary Completion 1994-12 (Actual); Study Completion 1994-12 (Actual)

PRIMARY OUTCOMES:
Benzodiazepine withdrawal severity

CONTACTS AND LOCATIONS:
Overall Officials: Scott Woods, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, Psychiatry, New Haven, Connecticut, United States

REFERENCES:
- [Background] Woods, et al., Soc Neuroscience Abstracts 21: 2098, 1995.